CLINICAL TRIAL: NCT04311229
Title: Effectiveness of Negative-Pressure Wound Therapy Compared to Wet-Dry Dressing in Pressure Injuries
Brief Title: Effectiveness of Negative-Pressure Wound Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20052020
Record Dates: First submitted 2020-02-28; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-02

CONDITIONS: Pressure Ulcers Stage III; Pressure Ulcer, Stage IV
Keywords: Negative-Pressure Wound Therapy; Pressure injuries; vacuum assisted closure; wound care; Wound Measurement
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: REPEATIVE MEASUREMENT EXPERİMENTAL AND CONTROL GROUPS
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative-Pressure Wound Therapy group (Experimental): NPWT was applied three times for Class III and pressure ulcers. An initial pre-treatment measurement was used as a baseline, followed by three post-treatment measurements after each round to evaluate wound healing. A total of four measurements were performed for each subject. Wound healing was measured using the PUSH Tool and the 3DWM device in both groups.
  Interventions: Device: Negative-Pressure Wound Therapy group
- CONTROL GROUP (Other): wet to dry dressing group
  Interventions: Other: contol group

INTERVENTIONS:
Device: Negative-Pressure Wound Therapy group — The wounds were initially evaluated for any necrotic findings and debrided if needed, and then washed with an antiseptic solution. 3-DWM was used to measure the pressure sores by taking pictures.The length and width of wounds were measured with disposable paper rulers. Wound depth was determined in centimeters with a sterile cotton-tip applicator by measuring against a ruler. The wound was closed using a Wound Care Kit that includes foam dressing, film drape, TRAC pad with tubing and a drainage canister. Foam material was placed inside the wound and was attached to the canister through tubing.The canister was attached to the Vacuum-Assisted Closure device, which is a portable device that applies intermittent or continuous negative pressure.The device was operated at 125 mmHg pressure for 5 minutes with and 2 minutes without active vacuum.Wound dressings were changed every 48 hours.Wound area was measured after all three rounds of treatment.
  Arms: Negative-Pressure Wound Therapy group
Other: contol group — Wounds were finally covered with gauze dressing soaked with saline. Wounds were treated three times a day, and measurements were repeated every 48 hours. Every wound was measured a total of four times: one pre-treatment (baseline) and three post-treatment measurements.
  Arms: CONTROL GROUP

SUMMARY:
This study aims to compare the effects of Negative-Pressure Wound Therapy and wet-to-dry dressing on Stages 3 and 4 pressure injuries, and to investigate the consistency of Three-Dimensional Wound Measurement Device findings with Pressure Ulcer Scale for Healing Tool scores. This study is a randomized controlled trial. A total of 30 patients with Stages 3 and 4 pressure injuries were included in the study. The patients were divided into two groups: the experimental group or Negative-Pressure Wound Therapy group and the control or wet-to-dry dressing group. All patients received 3 rounds of treatment. Data were collected with a Patient Identification Form, Pressure Ulcer Scale for Healing Tool and the findings of Three-Dimensional Wound Measurement Device. We found that granulation tissue formation was more significant in the experimental group (p < .05), and that there was more significant wound shrinkage (p < .05) with a more significant decrease in the Pressure Ulcer Scale for Healing Tool scores (p < .05). The wounds were assessed with the Tool and the Three-Dimensional Wound Measurement device. Device measurements were found to be correlated with Pressure Ulcer Scale for Healing Tool Tool findings (p < .05) There was a significant correlation between device-measured granulation findings and PUSH Tool score results of the experimental group's third measurements (p < .05). We conclude that Negative-Pressure Wound Therapy is an effective treatment method for pressure injuries, and Three-Dimensional Wound Measurement device is an usable wound assessment tool.

DETAILED DESCRIPTION:
Pressure injuries are a major health problem in that they are difficult to treat, reduce the patients' quality of life, and increase length of hospital stay and overall health care costs. Furthermore, several possible wound healing complications, such as infections, can lead to mortality. That said, the prevalence of pressure injuries is an important indicator of quality in hospitals. Pressure injuries do not only impact health, but also cause social isolation and dependency, resulting in further psychological problems.

Our review of the literature revealed that the incidence of pressure ulcers varies between 0.4% and 38% in hospitalized patients, between 2.2 and 23.9% in intensive care units and between 0-17% in home care. NPUAP (National Pressure Ulcer Advisory Panel) reports that the cost of treating pressure ulcers has been gradually increasing. It was estimated that treating pressure injuries costs around $11 billion annually in the United States alone. Treating a pressure ulcer can cost anywhere between $500 to $70,000, the most substantial fraction being nursing services. In the UK, it costs £1,064 to treat a Stage 1 pressure injury, and this number can reach £10,551 for more advanced ulcers. This illustrates the direct link between the stage of pressure injury and the cost of treatment. On average, it costs the UK healthcare system £1.4-2.1 billion annually to treat pressure ulcers.

There are many products and methods available for pressure ulcer treatment, but the most well-known and most commonly preferred method is wet-to-dry dressing. That said, researchers have tried and developed several novel methods for the treatment of pressure injuries including NPWT (Negative-Pressure Wound Therapy), hyperbaric oxygen therapy, ultrasonography, hydrotherapy, magnetic field therapy, ultraviolet rays, electrical stimulation, phototherapy and growth hormone application. Together with these non-invasive treatment methods, surgical intervention can also be a treatment option, especially for non-healing wounds. The European and US National Pressure Ulcer Advisory Panels' (EPUAP and NPUAP) guidelines recommend NPWT for deep-tissue pressure injuries, namely Stages 3 and 4, as a supportive tool for early-stage treatment. This method is based on applying negative pressure to promote wound healing. Several studies report that NPWT increases granulation tissue formation and reduces wound area. It is indicated that NPWT provides continuous and effective wound debridement in the wound area and increases blood supply to the wound.

Pressure injuries are among the most significant current health problems that are handled by a medical nurse. As the primary caregiver for the hospitalized patient, the nurse must prioritize preventing wound formation and eliminating any risk factors. If a pressure sore does form, the primary goal is to plan and implement appropriate care and nursing interventions in collaboration with the patient and their family to ensure proper wound healing .

It is the nurse's responsibility to keep up with scientific developments in patient care and try to integrate them into their work. PUSH is a tool that is used for monitoring pressure ulcers; however, it has yet to become a part of routine practice in Turkey. The Three-Dimensional Wound Management (3-DWM) device has been used in medical service since 2015, but with only a limited number of studies that evaluate its effectiveness. Currently, the wet-to-dry dressing method is the most commonly preferred treatment method for wound care in Turkish healthcare. There are indeed numerous studies that demonstrate the effectiveness of wet dressings in wound healing. Wet dressings provide the appropriate medium for the accumulation of patient's own body fluids between wound surface and dressing while preventing dehydration. This study aims to compare the effects of Negative-Pressure Wound Therapy (NPWT) and wet-to-dry dressing on Stages 3 and 4 pressure injuries, and to investigate the consistency of 3-DWM device measurement findings with PUSH Tool scores.

ELIGIBILITY:
Inclusion Criteria:

* having class III or IV pressure ulcer
* being ≥18 years old,
* not having time/access constraints,
* voluntariness.

Exclusion Criteria:

* Stage I and Stage II pressure ulcers,
* cancer,
* increased risk of bleeding,
* osteomyelitis,
* corticosteroid treatment
* consciousness and
* contraindications of NPWT

Ages: 18 Years to 79 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Granulation tissue formation and wound shrinkage | 8 week
  Granulation tissue formation (%) and wound shrinkage (cm²) in experimental and control groups
PUSH tool and 3-DWM measurement findings | 8 week
  Wound area assessed by PUSH tool and wound area and granulation tissue assessed by 3-DWM device

CONTACTS AND LOCATIONS:
Overall Officials: EZGİ ARAYAN, Msc, Principal Investigator — BAŞKENT ÜNİVERSİTESİ İSTANBUL SAĞLIK UYGULAMA VE RAŞTIRMA MERKEZİ; SELDA RIZALAR, Assoc.Prof., Study Director — İSTANBUL MEDİPOL ÜNİVERSİTESİ; EMRE ÖZKER, Assoc.Prof., Study Director — BAŞKENT ÜNİVERSİTESİ İSTANBUL SAĞLIK UYGULAMA VE RAŞTIRMA MERKEZİ

IPD SHARING:
Plan to Share IPD: Yes
to publish the article
Supporting Information: Study Protocol
Time Frame: 2020
Access Criteria: all academician and practicioners

REFERENCES:
- [Background] Ersilia LA, Anagha K, Thomas EB, KAthryn MM, John SS, Karen KE, Paul JK, Christopher EA, Reliability of a novel 3D Wound Measurement Device, 2015
- [Background] Bills JD, Berriman SJ, Noble DL, Lavery LA, Davis KE. Pilot study to evaluate a novel three-dimensional wound measurement device. Int Wound J. 2016 Dec;13(6):1372-1377. doi: 10.1111/iwj.12534. Epub 2015 Nov 11. PMID 26558349
- [Background] Moues CM, van den Bemd GJ, Heule F, Hovius SE. Comparing conventional gauze therapy to vacuum-assisted closure wound therapy: a prospective randomised trial. J Plast Reconstr Aesthet Surg. 2007;60(6):672-81. doi: 10.1016/j.bjps.2006.01.041. Epub 2006 Jun 22. PMID 17485058
- [Background] Sinha K, Chauhan VD, Maheshwari R, Chauhan N, Rajan M, Agrawal A. Vacuum Assisted Closure Therapy versus Standard Wound Therapy for Open Musculoskeletal Injuries. Adv Orthop. 2013;2013:245940. doi: 10.1155/2013/245940. Epub 2013 Jun 26. PMID 23878741
- See also: National Pressure Ulcer Advisory Panel — https://npiap.com/default.aspx
- See also: NPUAP (NationalPressureUlcerAdvisory Panel). "Prevention and Treatment of Pressure Ulcers: Quick Reference Guide". — https://www.epuap.org/wp-content/uploads/2010/10/Quick-Reference-Guide-DIGITAL-NPUAP-EPUAP-PPPIA-16Oct2014.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04311229/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04311229/ICF_001.pdf